CLINICAL TRIAL: NCT06863441
Title: The Value of PET Imaging Targeting Granzyme B in Predicting Efficacy and Prognosis in T-NK Cell Lymphoma
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, LI BIAO, chief physician, Ruijin Hospital
Other Study IDs: RuijinH 2025-34
Record Dates: First submitted 2025-02-20; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: T-NK Cell Lymphoma
Keywords: PET/CT; Granzyme B; immunotherapy
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients diagnosed with T-NK cell lymphoma who will receive immunotherapy

SUMMARY:
The study on the value of PET imaging targeting granzyme B in predicting the efficacy and prognosis of T-NK cell lymphoma.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo 68Ga-grazytracer PET at baseline and after one course of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years, regardless of gender.
2. Histopathologically confirmed diagnosis of T-NK cell lymphoma.
3. Newly diagnosed and untreated patients or refractory/relapsed patients preparing to undergo immunotherapy.
4. Availability of complete clinicopathological and follow-up data.
5. Signed and dated informed consent form.

Exclusion Criteria:

1. Patients who have previously received anti-tumor therapy.
2. Patients with a history of other malignancies.
3. Incomplete clinical information or imaging data.
4. Concurrent other malignant tumors.
5. Patients with severe medical conditions deemed unsuitable for participation in this clinical study by the investigator, such as severe cardiopulmonary insufficiency or severe hepatic and renal dysfunction.
6. Poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patient with pathologically confirmed T-NK cell lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | Baseline and 7-10 days after treatment
  SUV of 68Ga-grazytracer uptake on PET/CT images for tumor lesions

SECONDARY OUTCOMES:
Progress free suivival | 3 years
  Progress free suivival
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University Medical School, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No